CLINICAL TRIAL: NCT00836875
Title: A Prospective, Open-label, Non-randomized, Multi-center Study To Investigate The Safety And Tolerability Of Voriconazole As Primary Therapy For Treatment Of Invasive Aspergillosis And Molds Such As Scedosporium Or Fusarium Species In Pediatric Patients.
Brief Title: A Study To Evaluate The Safety Of Voriconazole As Treatment Of Invasive Aspergillosis (Fungal Infection) And Other Rare Molds In Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This protocol terminated prematurely on July 8, 2013 due to slow enrollment, not because of any safety issues or concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A1501080; 2008-005275-10 (EudraCT Number)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Invasive Aspergillosis
Keywords: Pediatrics voriconazole invasive fungal infection invasive aspergillosis immunocompromized
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Children from 2 to 17 years who have possible, probable or proven invasive aspergillosis, or other rare mold infection (eg, Scedosporium and Fusarium).
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — All subjects will receive voriconazole for a minimum of 6 weeks and a maximum of 12 weeks. All subjects must receive intravenous (IV) voriconazole for the first week of therapy.
  Group 1: Subjects 2 to 11 years old and subjects 12 to 14 years old with low body weight (<50 kg) will receive 9 mg/kg IV every 12 hours (q12h) on day 1, then 8 mg/kg IV q12h starting day 2. If there is a significant clinical improvement after the first week of IV therapy, subjects may be switched to the step-down oral regimen (9 mg/kg PO q12h with a maximum dose of 350 mg PO q12h) at the discretion of the investigator.
  Group 2: Subjects 12 to 17 years old (excluding 12-14-year-olds weighing <50 kg) will receive 6 mg/kg IV q12h on day 1, then 4 mg/kg IV q12h starting day 2. Similar to Group 1, subjects may be switched to the step-down oral regimen (200 mg PO q12h) at the discretion of the investigator. Oral voriconazole can be administered as tablet or oral suspension.

SUMMARY:
The purpose of this study is to evaluate the safety profile of voriconazole (an antifungal drug) when used in children who have invasive aspergillosis (IA) and other rare systemic fungal infections.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised with clinically compatible illness.
* Diagnosis of proven or probable or possible Invasive Aspergillosis (based on a modified version of the revised EORTC/MSG consensus definitions).
* Diagnosis of infection due to Scedosporium or Fusarium species.
* Male and female from 2 to 17 years of age.
* Females with childbearing potential must have negative pregnancy test and be using appropriate contraception.

Exclusion Criteria:

* Allergy or hypersensitivity to the azole drugs.
* Female subjects who are pregnant or lactating.
* Patients who received more than four days of antifungal drugs to treat the current episode of invasive aspergillosis or rare mold infection.
* Received within 24 hours prior to enrollment drugs that may cause QT interval prolongation.
* Significant liver, kidney or heart dysfunction.
* Not expected to survive for at least 5 days.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (9):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center Oakland (CHRCO), Oakland, California
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Children's Pavilion, Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Commonwealth University Health System, Hospital Pharmacy, Richmond, Virginia
  - Pediatric Hematology and Oncology, Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Commonwealth University/MCV Clinical Pathology, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - Alberta Children's Hospital, Pediatric Oncology Office, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
- Fakultni nemocnice Brno, Brno, Czechia
- UMC St. Radboud, Nijmegen, Netherlands
- Klinika Transplantacji Szpiku, Onkologii i Hematologii Dzieciecej, Wroclaw, Poland
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- Spain (5):
  - Hospital General Universitari Vall D'Hebron, Barcelona
  - Hospital Universitari Vall d'Hebron. Servicio de Farmacia, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - HOSPITAL UNIVERSITARIO 12 DE OCTUBRE Servicio de Farmacia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Thailand (3):
  - Department of Pediatrics, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Department of Pediatrics, Faculty of Medicine, Chulalongkorn University, Patumwan, Bangkok
  - Department of Pediatrics, Phramongkutklao hospital, Rajathevee, Bangkok

REFERENCES:
- [Derived] Martin JM, Macias-Parra M, Mudry P, Conte U, Yan JL, Liu P, Capparella MR, Aram JA. Safety, Efficacy, and Exposure-Response of Voriconazole in Pediatric Patients With Invasive Aspergillosis, Invasive Candidiasis or Esophageal Candidiasis. Pediatr Infect Dis J. 2017 Jan;36(1):e1-e13. doi: 10.1097/INF.0000000000001339. PMID 27636722
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501080&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20Of%20Voriconazole%20As%20Treatment%20Of%20Invasive%20Aspergillosis%20%28Fungal%20Infection%29%20And%20Other%20Rare%20Molds%20In%20C

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole: 2 to <12 Years: Participants aged 2 to less than (<)12 years (and young adolescents aged 12 to 14 years weighing <50 kilograms [kg]) received a loading dose of voriconazole of 9 milligrams per kg (mg/kg), intravenously (IV), every 12 hours (q12h) for the first 24 hours, followed by maintenance dosing of 8 mg/kg IV q12h for a minimum of 7 days of IV therapy. Once significant clinical improvement was observed, participants could have been switched or oral (PO) therapy and received 9 mg/kg PO voriconazole q12h for a maximum dose of 350 mg.
- Voriconazole: 12 to <18 Years: Participants aged 12 to <18 years (excluding those aged 12-14 years weighing <50 kg) received a loading dose of 6 mg/kg IV q12h for the first 24 hours followed by maintenance dosing of 4 mg/kg IV q12h for a minimum of 7 days of IV therapy. Once significant clinical improvement was observed, participants could have been switched or oral therapy and received 200-300 mg PO q12h.
Period: Overall Study
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Started | 11 | 20
Completed | 8 | 17
Not Completed | 3 | 3
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years | Total
Number analyzed (Participants) | 11 | 20 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (2.3) | 14.1 (1.7) | 11.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Baseline, daily while hospitalized, Days 7, 14, 28, 42, 84, and 114, at end of treatment, and up to 1 month post treatment
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 11 | 20
participants
  With AEs | 11 | 19
  With serious AEs | 6 | 9
  With severe AEs | 5 | 8
  Discontinued treatment due to AEs | 1 | 0
  Dose reduced or temporarily discontinued due to AE | 0 | 4

2. Secondary Outcome: Percentage of Participants With a Global Response of Success
Description: Percentage of participants with global response of success at Weeks 6 and at EOT (up to Week 12). Global response of success was defined as a participant who achieved a complete or partial global response per the investigator. Complete response was defined as resolution of all clinical signs and symptoms PLUS resolution of 90 percent (%) or more of the lesions visible on radiological studies and attributed to invasive aspergillosis (IA) at Baseline. Partial response was defined as clinical improvement PLUS 50% to <90% resolution of the radiological lesions attributed to IA at Baseline.
Time Frame: Weeks 6 and End of Treatment (EOT; up to Week 12)
Population: Modified intent to treat (MITT) population: all participants receiving at least 1 dose of study drug and diagnosed with proven or probable aspergillosis (defined by modified European Organization for Research and Treatment of Cancer Mycoses Study Group [EORTC/MSC] criteria) or microbiologically confirmed scedosporium or fusarium infection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 5 | 9
percentage of participants
  Week 6 | 40.0 [5.3 to 85.3] | 77.8 [40.0 to 97.2]
  EOT | 40.0 [5.3 to 85.3] | 77.8 [40.0 to 97.2]

3. Secondary Outcome: All-Cause Mortality - Number of Participant Deaths
Description: Number of participant deaths reported at Week 6 and at EOT (up to Week 12).
Time Frame: Week 6 and EOT (up to Week 12)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 11 | 20
participants
  Week 6 | 3 | 1
  EOT | 0 | 1

4. Secondary Outcome: Attributable Mortality - Number of Participant Deaths
Description: Number of participant deaths attributable to study drug reported at Week 6 and at EOT (up to Week 12).
Time Frame: Weeks 6 and EOT (up to Week 12)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 11 | 20
participants | 0 | 0

5. Secondary Outcome: Time to Death
Time Frame: Baseline up to 1 month post treatment
Population: Safety population; only participants who died were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 3 | 2
days | 30.0 [18 to 38] | 47.5 [20 to 75]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Serious Adverse Events (participants affected / at risk) | 6/11 | 9/20
Other Adverse Events (participants affected / at risk) | 10/11 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole: 2 to <12 Years (N=11) | Voriconazole: 12 to <18 Years (N=20)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Aspergillosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endotracheal intubation (Surgical and medical procedures) | 0 | 1
Aneurysm ruptured (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole: 2 to <12 Years (N=11) | Voriconazole: 12 to <18 Years (N=20)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1
Asthenopia (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Chromatopsia (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 2
Diplopia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 3
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Painful defaecation (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Catheter site discharge (General disorders) | 0 | 1
Catheter site pain (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 7
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Implant site pustules (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Incorrect drug administration rate (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 2
Oxygen saturation decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Respirovirus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 2
Lethargy (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Genital swelling (Reproductive system and breast disorders) | 1 | 0
Vulvar erosion (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to slow enrollment. The study was not terminated due to any safety issues or concerns. Interpretation of the data are limited due to the small sample size and descriptive design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.